CLINICAL TRIAL: NCT00973115
Title: Efficacy and Safety of Morning Versus Evening Intake of Simvast CR Tablet in Patients With Hyperlipidemia: A Randomized, Double-blind, Multicenter Phase 3 Trial
Brief Title: Efficacy and Safety of Morning Versus Evening Intake of Simvast Controlled Release (CR) Tablet in Patients With Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HM-SIM-302
Record Dates: First submitted 2009-09-06; First posted 2009-09-09 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Hyperlipidemia
MeSH Terms: conditions — Hyperlipidemias

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simvastatin CR 20mg- morning administration (Experimental)
  Interventions: Drug: Simvastatin CR
- Simvastatin CR 20mg- evening administration (Active Comparator)
  Interventions: Drug: Simvastatin CR

INTERVENTIONS:
Drug: Simvastatin CR

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of morning versus evening intake of Simvastatin Controlled Release tablet 20mg for 8 weeks in patients with hyperlipidemia. This study will investigate equivalence of the low-density lipoprotein(LDL) cholesterol percent change.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 19 and 75
* Defined as a fasting 100mg/dl≤ LDL cholesterol <220mg/dl and triglyceride level<400 mg/dl
* Need drug therapy by NCEP ATP III guideline
* Signed informed consent

Exclusion Criteria:

* Has a hypersensitivity to HMG-CoA reductase inhibitor or simvastatin
* Has a presence or history of alcohol abuse or drug abuse
* Active gallbladder disease within 12 months
* Pancreatitis or Hepatic dysfunction (ALT or AST levels > 2XUNL)
* HbA1c≥ 9% in type 2 diabetes mellitus patients
* SBP < 90mmHg or > 160mmHg
* DBP < 50mmHg or > 100mmHg
* Myocardial infarction or revascularization procedure within 6 months
* Has significant cardiovascular disease
* Malignant tumor within 5years
* Has fibromyalgia, myopathy, rhabdomyolysis or acute myalgia
* Uric acid level > 9 mg/dl
* Thyroid stimulating hormone ≥ 2XUNL
* Active peptic ulcer disease
* CPK levels > 3XUNL
* creatinine level > 2 mg/dl
* Negative pregnancy test for women of childbearing age and agreement to use contraception while on study
* Had participated other clinical trial within 4 weeks
* Need systemic administration of corticosteroids intermittently

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2007-11; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
the percent change from baseline in LDL cholesterol | week 8

SECONDARY OUTCOMES:
the change and the percent change from baseline for total cholesterol, HDL cholesterol, Triglyceride, apolipoprotein A-I, apolipoprotein B, and lipoprotein(a) | week 8

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hoon Park, M.D., Ph.D, Principal Investigator — Ehwa Womans University Mokdong Hospital
Locations (1):
- 8 Sites, Seoul, South Korea